CLINICAL TRIAL: NCT04031625
Title: Prospective and Retrospective Metastatic Colorectal Cancer Database
Brief Title: Metastatic Colorectal Cancer Database
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: AB2012CR
Record Dates: First submitted 2019-07-01; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic Colorectal Cancer
  Interventions: Other: Metastatic Colorectal Cancer Database

INTERVENTIONS:
Other: Metastatic Colorectal Cancer Database — Metastatic Colorectal Cancer Database

SUMMARY:
The metastatic ColoRectal Cancer (mCRC) Database base contains data collected during the regular clinical patient management in Centre Georges Francois Leclerc, Dijon.

DETAILED DESCRIPTION:
The metastatic ColoRectal Cancer (mCRC) Database base contains data collected during the regular clinical patient management (sociodemographic, clinical, pathological, radiological, biological, disease evolution, ...). This database allows easy access to information in a centralized and structured way. This cohort is used to gather insights for research purposes.

All data collected come from medical files of patients managed at Centre Georges Francois Leclerc, Dijon, France.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer
* Age >= 18

Exclusion Criteria:

* Non metastatic colorectal cancer
* Objection to the use of medical data records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Regular clinical metastatic colorectal patient management in Centre Georges François Leclerc, Dijon
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-11-26 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Patient survival | 2 years
  Overall survival and evolution over years

SECONDARY OUTCOMES:
Collection of patient and treatment characteristics | 2 years
  Collection of patient and treatment characteristics over years, to set up prospective and retrospective studies

CONTACTS AND LOCATIONS:
Locations (1):
- Methodology, Biostatistics and Data Management, Dijon, France

IPD SHARING:
Plan to Share IPD: No